CLINICAL TRIAL: NCT02910947
Title: Comparative Evaluation of Quadratus Lumborum and Transverses Abdominis Plane Block for Postoperative Pain Relief in Lower Abdominal Surgeries
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr Vikas Saini, Associate professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: INT/IEC/2016/2146
Record Dates: First submitted 2016-09-16; First posted 2016-09-22 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Pain Relief to the Patient Following Abdominal Surgeries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- quadratus lumborum (Experimental)
  Interventions: Procedure: ultrasound guided quadratus lumborum or Transversus Abdominis plane block
- TAP(Transversus abdominis plane) (Experimental)
  Interventions: Procedure: ultrasound guided quadratus lumborum or Transversus Abdominis plane block

INTERVENTIONS:
Procedure: ultrasound guided quadratus lumborum or Transversus Abdominis plane block — The intervention consists of giving ultrasound guided local anaesthetic (0.125% bupivacaine ) in the quadratus lumborum plane or the transversus abdominis plane after randomization. These planes and technique for these procedures are well described in literature.

SUMMARY:
Two ultrasound guided techniques to give postoperative pain relief to the patients following abdominal surgeries would be compared using scoring systems for pain relief and scientific methods. while one technique is routinely used, other i.e quadratus lumborum has been recently described and relies on posterior deposition of the drug. Both the techniques are safe and ultrasound imaging is to be used for guidance.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing lower abdominal surgery 18-60 yrs of age

Exclusion Criteria:

* none

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
pain relief following abdominal surgery. Visual Analogue Scale (VAS) would be used to record pain at rest. In this patient is asked to describe his/her pain on a scale from 0-10. | 24 hrs

CONTACTS AND LOCATIONS:
Locations (1):
- PGIMER, Chandigarh, Chandigarh, India